CLINICAL TRIAL: NCT03365661
Title: QUILT-3.034: Multi-Center Trial of Non-Myeloablative TCRa/b Deplete Haploidentical Hematopoietic Cell Transplantation With Post HCT ALT-803 in High-Risk Myeloid Diseases
Brief Title: QUILT-3.034: Non-Myeloablative TCRa/b Deplete Haplo HSCT With Post ALT-803 for AML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor halted study.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS057; MT2016-06 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2017-12-03; First posted 2017-12-07 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: High-Risk Acute Myeloid Leukemia; Treatment-Related Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALT-803 (Experimental)
  Interventions: Biological: ALT-803

INTERVENTIONS:
Biological: ALT-803 — A reduced intensity conditioning starts on Day -6, (CY/FLU/TBI/TLI) followed by infusion of a TCRα/β-deplete haploidentical graft on Day 0. Two doses of ALT-803 are given initially (early) 1 week apart to facilitate NK cell expansion. ALT-803 maintenance (late) for immune reconstitution begins at Day 42 and consists of 4 weekly doses, followed by 4 weeks off. Up to four 8 week treatment courses are permitted. No post-transplant GVHD prophylaxis is administered unless the final donor cell product contains > 2 x 105 α/β T cells/kg recipient weight.

SUMMARY:
This is a phase II multi-institutional therapeutic study of a non-myeloablative T cell receptor (TCR) alpha/beta depleted haploidentical transplantation with post-transplant immune reconstitution using ALT-803 for the treatment of high-risk myeloid leukemia (AML), treatment-related/secondary AML, and myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to ≤70 years
* Meets one of the following disease and risk categories:

  * High-Risk Acute Myeloid Leukemia (AML) with predicted risk of relapse higher than 30%, which includes, but not limited to the following:

    * Patients in morphological remission (CR1 or beyond) with minimal residual disease as quantified either by flow cytometry, or by cytogenetics or molecular markers.
    * Patients with the following karyotypes in morphological CR or CRi: ELN-Intermediate I, Adverse, ELN-Intermediate-II. (18) (Examples include monosomal karyotype, complex karyotype, mutant p53, mutant RUNX1, mutant ASXL1, mutant FLT3-ITD, mutant DNMT3A, Inversion 3, T(6:9), KIT mutated core binding factor AML)
  * Treatment-Related AML and Secondary AML in morphological remission (CR1 or beyond) with minimal residual disease as quantified either by flow cytometry, or by cytogenetics or molecular markers
  * Myelodysplastic Syndrome (MDS) with < 5% blasts by morphology and meets at least one of the following:

    * Received intensive induction chemotherapy (i.e. 7+3 or MEC) OR
    * Progression after 4 cycles of hypomethylating agents
  * The donor and recipient must be HLA identical for at least one haplotype (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1
* Karnofsky performance status ≥ 60% (appendix IV)
* Adequate organ function within 14 days of study registration (30 days for pulmonary and cardiac) defined as:

  * Hepatic: AST and ALT < 3 x upper limit of institutional normal
  * Renal: estimated glomerular filtration rate (GFR) ≥ 40 mL/min/1.73m2
  * Pulmonary: oxygen saturation ≥ 90% on room air with no symptomatic pulmonary disease. If symptomatic or prior known impairment DLCOcor ≥ 40%.
  * Cardiac: LVEF ≥ 40% by echocardiography, MUGA, or cardiac MRI, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to transplant (excluding preparative regimen pre-medications)
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

* Acute leukemias of ambiguous lineage
* Allogeneic transplant for AML within the previous 6 months (no time limit for autologous transplant)
* Active CNS disease - if a history of AML related CNS involvement, screening CSF analysis must be negative
* Pregnant or breastfeeding - The agents used in this study include those that fall under Pregnancy Category D - have known teratogenic potential. Women of child bearing potential must have a negative pregnancy test at screening
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on systemic chronic medications (mild asthma requiring inhaled steroids only is eligible)
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections including HIV-1/2 or active hepatitis C/B - chronic asymptomatic viral hepatitis is allowed
* Active concomitant second malignancy (i.e. has required treatment in the previous 6 months)
* Known hypersensitivity to any of the study agents
* Received any investigational drugs within the 14 days before 1st dose of fludarabine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of disease response | Day 28
  Rate of donor neutrophil engraftment in the absence of disease at Day +28. Neutrophil engraftment is defined as absolute neutrophil count (ANC) ≥ 5 X 10 8 /L.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 12 months
  Incidence of disease free survival (DFS).
Treatment Related Mortality (TRM) | 12 months
  Incidence of treatment related mortality (TRM).
Disease Relapse | 12 months
  Incidence of disease relapse.
Grade II-IV acute Graft versus Host Disease (aGVHD) | Day 100
  Incidence of acute Graft versus Host Disease measured by the number of T-cells infused or NK cells engrafted causing GVHD syndrome.
Serious Adverse Events from ALT-803 (Early Schedule) | 1 Year
  Incidence of serious adverse events from ALT-803 will be measured for an initial 2 doses, given one week apart.
Serious Adverse Events from ALT-803 (Late Schedule) | 1 Year
  Incidence of serious adverse events from ALT-803 will be measured for 16 doses, given over 4 weeks.
Chronic Graft versus Host Disease (cGVHD) | 1 year
  Incidence of chronic Graft versus Host Disease will be measured by the number of T-cells infused or NK cells engrafted causing GVHD syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cooley, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States